CLINICAL TRIAL: NCT07038551
Title: Prophylactic Use of Naldemedine on Opioid-Induced Nausea and Vomiting in Patients With Cancer: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Prophylactic Use of Naldemedine on Opioid-induced Nausea and Vomiting in Patients With Cancer: POSEIDON Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: International University of Health and Welfare (Other)
Collaborators: Shionogi (Industry)
Responsible Party: Principal Investigator, Takaomi Kessoku, M.D., Ph.D., International University of Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024U0160
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Opioid-Induced Constipation (OIC)
Keywords: Nausea; Vomiting; Constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Nausea; Vomiting; Constipation | interventions — naldemedine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naldemedine (Active Comparator)
  Interventions: Drug: Naldemedine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naldemedine — over-encapsulated capsule of either 0.2 mg of naldemedine
  Arms: Naldemedine
Drug: Placebo — over-encapsulated capsule of placebo
  Arms: Placebo

SUMMARY:
Opioid analgesics can cause side effects such as constipation, nausea, and vomiting by acting on opioid receptors widely distributed in the peripheral nervous system. This can sometimes make it difficult to achieve and maintain pain relief and continue pain treatment. Among these side effects, nausea and vomiting are specifically referred to as opioid-induced nausea and vomiting (OINV). OINV is known to occur during the initial administration or dose escalation of opioid analgesics, and it not only decreases the quality of life for patients but also reduces adherence to opioid analgesics, which can have a negative impact on pain management. Therefore, appropriate management is crucial.

While the administration of conventional antiemetic drugs is recommended for the treatment of OINV, there is a lack of high-quality studies evaluating their effectiveness, and studies comparing treatment effects with a placebo have not been reported.

The objective is to verify the effectiveness of nalbuphine in preventing OINV in patients starting opioid analgesics for cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can be expected to initiate regular administration of opioid analgesics (tramadol, morphine, oxycodone, hydromorphone) for cancer pain and continue for 7 days or more.
2. Patients who are 18 years of age or older at the time of obtaining consent
3. Patients who can take oral medications, food, and beverages
4. Patients who are considered capable of self-recording in the patient's diary (proxy recording in the patient's diary is acceptable if the patients are capable of self-assessment).
5. Patients who are not expected to have a rapid change in their condition during the study period.
6. Patients who can obtain written consent to participate in the study of their own will

Exclusion Criteria:

1. Patients who have used opioid analgesics within 28 days prior to the date of consent
2. Patients who have taken or are currently taking naldemedine
3. Patients who have nausea and vomiting of CTCAE grade 2 or higher at the time of obtaining consent
4. Patients who have taken the following antiemetic drugs within 7 days prior to the date of consent Metoclopramide, domperidone, H1 histamine receptor antagonists, phenothiazine antipsychotics (chlorpromazine, levomepromazine, prochlorperazine), haloperidol, atypical antipsychotics (perospirone, risperidone, olanzapine), serotonin 5HT3 receptor antagonists (ondansetron, granisetron, ramosetron, palonosetron), corticosteroids (dexamethasone), scopolamine hydrobromide, NK1 receptor antagonists (aprepitant, fosaprepitant, fosnetupitant)
5. Patients who have received cancer chemotherapy that is certain to affect nausea and vomiting within 14 days prior to the initial enrollment date, or who are scheduled to receive such therapy within the study period. Cancer chemotherapy that is certain to affect nausea and vomiting will be defined as follows:

   ① Initial administration of a therapeutic regimen containing irinotecan (CPT-11)

   ② Other cancer chemotherapy that is considered certain to affect nausea and vomiting.

   However, the following cases may be considered as not affecting defecation
   * Chemotherapy with the same regimen as the previous course or chemotherapy with the same drug and dose, and there was no moderate or greater nausea and vomiting (CTCAE v5.0 Grade 2 or higher) during the previous course or previous chemotherapy.
   * Patients who have received oral anticancer agents (e.g. TS-1) daily and have not had moderate or severe nausea and vomiting (CTCAE v5.0 Grade 2 or higher) for at least 1 week from the start of oral chemotherapy to the start of study drug.
6. Pregnant or lactating patients
7. Patients with suspected hypersensitivity to opioid receptor antagonists such as naldemedine, naltrexone, methylnaltrexone, and naloxone
8. Patients with contraindications listed in the package inserts for naldemedine and opioid analgesics (tramadol, morphine, oxycodone, hydromorphone)
9. Patients participating or scheduled to participate in clinical trials or other interventional studies
10. Patients with gastrointestinal obstruction or suspected gastrointestinal obstruction, or patients with a history of gastrointestinal obstruction and a high risk of recurrence
11. Patients who have undergone surgery or treatment (e.g., nerve block) that affects gastrointestinal function, or radiation therapy to the head, abdomen, or pelvis within 14 days prior to the date of consent acquisition, or patients who are scheduled to undergo such treatment during the observation period
12. Patients with medically significant cardiovascular, respiratory, hepatic, or renal dysfunction based on history, clinical laboratory values, electrocardiogram, or physical examination, who are judged inappropriate to participate in the study
13. Patients with symptomatic intracranial conditions (such as brain metastases or leptomeningeal disease)
14. Patients with suspected dysfunction or impairment of the blood-brain barrier
15. Patients for whom it is difficult to explain the contents of the study or obtain consent due to cognitive impairment or psychiatric illness
16. Patients who are judged by the principal investigator or sub-investigator to be inappropriate to participate in this study based on other concomitant therapies or medical findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved a Complete Response on Day 5 (CR5), defined as no vomiting up to 120 hours after starting opioid analgesic and no use of rescue antiemetic medications. | 120 hours

SECONDARY OUTCOMES:
The proportion of patients who achieved a Complete Response at CR1, CR2, CR3, and CR7 (defined as no vomiting up to 24, 48, 72, and 168 hours after starting opioid analgesics, respectively, and no use of rescue antiemetic medications) | 24, 48, 72, and 168 hours
Change in nausea NRS from baseline | Day 1, 2, 3, 5, and 7
  nausea NRS[0-10]: Higher scores indicate greater nausea intensity
Average duration of nausea per day | Day 1, 2, 3, 5, and 7
Proportion of patients who vomited at least once after starting opioid analgesics | 24, 48, 72, 120, and 168 hours
Proportion of patients who used rescue antiemetic medicines | 24, 48, 72, 120, and 168 hours
Number of times rescue antiemetic medicines were used | 24, 48, 72, 120, and 168 hours
Proportion of patients with Spontaneous Bowel Movement (SBM: spontaneous bowel movement) of 3 or more per week | 7days
Proportion of patients with Spontaneous Bowel Movement (CSBM: SBM without residual defecation) of 3 or more per week | 7days
Proportion of patients experiencing a sensation of residual defecation in 25% or more of defecation | 7days
Proportion of patients with SBM without urgency of 3 or more per week | 7days
Proportion of patients experiencing a sensation of urgency in 25% or more of defecation | 7days
Proportion of patients with SBM without urgency or residual defecation of 3 or more per week | 7days
Proportion of patients experiencing a sensation of urgency or residual defecation in 25% or more of defecation | 7days
Number of times rescue laxatives or enema or digital evacuation were used | 7days
Proportion of patients with a Bowel Function Index of less than 28.8 | 7days
Change in Bowel Function Index from baseline | 7-11days
the percentage of patients whose satisfaction worsened | 7-11days
Change in Global Quality of Life score and scores for each subscale evaluation of the EORTC-QLQ-C15 PAL | 7-11days
Change in pain NRS from baseline | 1,2,3,5,7days
  pain NRS[0-10]: Higher scores indicate greater pain intensity

CONTACTS AND LOCATIONS:
Locations (1):
- International university of health and welfare Narita hospital, Narita, Japan